CLINICAL TRIAL: NCT05501743
Title: Evaluation of the Efficacy of an Intra-articular Injection of Autologous Microfat Combined With Autologous Platelet-enriched Plasma in the Treatment of Radiocarpal Osteoarthritis: a Randomized Controlled Non-inferiority Trial Versus Total Wrist Denervation.
Brief Title: Evaluation of the Efficacy of an Intra-articular Injection of Autologous Microfat Combined With Autologous Platelet-enriched Plasma in the Treatment of Radiocarpal Osteoarthritis: a Randomized Controlled Non-inferiority Trial Versus Total Wrist Denervation (Established Standard Treatment).
Acronym: AMIPREP-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-006817-12
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Arthrosis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Randomization will be balanced in 2 parallel groups :
  * Patients in the "study treatment" group (T) will receive an intra-articular injection of microfat and PRP.
  * Patients in the "reference treatment" group (R) will undergo total wrist denervation surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study treatment group (T) (Experimental): The treatment by intra-articular injection of autologous microfat and PRP will be performed during a half-day outpatient stay in the hand and limb repair surgery department at the Hôpital de la Timone. The total duration of the procedure is approximately 4 hours and includes 2 surgical times performed in the operating room and an intermediate waiting time for the patient in an outpatient room during the preparation of the experimental products.
  Interventions: Drug: Intra-articular injection of microfat and PRP
- Reference treatment group (R) (Active Comparator): The surgical treatment by total denervation of the wrist will be performed during a one-day outpatient stay in the hand and limb surgery department at the Hôpital de la Timone. It will be performed under loco-regional anesthesia by axillary plexus block.
  Interventions: Procedure: Total denervation of the wrist

INTERVENTIONS:
Drug: Intra-articular injection of microfat and PRP — The treatment by intra-articular injection of autologous microfat and PRP will be performed during a half-day outpatient stay in the hand and limb repair surgery department at the Hôpital de la Timone. The total duration of the procedure is approximately 4 hours and includes 2 surgical times performed in the operating room and an intermediate waiting time for the patient in an outpatient room during the preparation of the experimental products.
  Arms: Study treatment group (T)
Procedure: Total denervation of the wrist — The surgical treatment by total denervation of the wrist will be performed during a one-day outpatient stay in the hand and limb surgery department at the Hôpital de la Timone. It will be performed under loco-regional anesthesia by axillary plexus block.
  Arms: Reference treatment group (R)

SUMMARY:
This is a phase II, prospective, comparative, randomized, single-center, open-label, parallel-group therapeutic trial.

It is a non-inferiority trial to establish the efficacy of intra-articular injection of autologous microfat and PRP at the wrist in patients suffering from radiocarpal osteoarthritis in reference to wrist denervation.

DETAILED DESCRIPTION:
The main objective is to demonstrate the non-inferiority of the efficacy of intra-articular injection of autologous microfat and PRP in patients suffering from radiocarpal osteoarthritis resistant to medical treatment on pain evaluated by the visual analog scale (VAS) at 6 months in comparison with total denervation of the wrist (reference treatment).

Secondary objectives are:

* To assess the safety of the study treatment at D7, M3, M6, M12, compared to the reference treatment group: Adverse events and post-operative follow-up data.
* To assess the non-inferiority of the study treatment compared to the reference treatment on the secondary efficacy criteria.
* Evaluate the effectiveness of the treatment under study.
* Evaluate patient satisfaction.
* To investigate the existence of a relationship between the characteristics of the injected products and the clinical improvement and to describe the characteristics of the responder and non-responder patients. The responder patient was characterized by an improvement of the VAS at 6 months superior to the minimal clinically significant difference fixed at 14 points.
* To evaluate the improvement of cartilage relaxation time on high-resolution T2 gradient echo and Turbo Spin Echo 3T MRI sequences at 6 months in patients in the "study treatment" group.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged ≥ 18 years
* Patients with wrist osteoarthritis:
* Symptomatic: pain ≥ 40 mm on the visual analog scale (VAS 0-100 mm) more or less associated with a loss of strength objectified by the Jamar dynamometer and/or wrist mobility leading to discomfort in activities of daily living and impaired quality of life.
* Objectivated on radiographs and arthroscanner: stylo-scaphoid and/or global radiocarpal and/or scapho-capital and/or luno-capital joint pinch, more or less associated with osteophytic and subchondral changes equivalent to a grade 3 of the Kellgren and Lawrence classification (see chapter I). Depending on the etiology of the wrist osteoarthritis, the following may be associated: an adaptive carpal defect (DISI), a rupture of the scapholunate or pisotiquetral ligaments, a pseudarthrosis of the scaphoid, a necrosis of the proximal pole of the scaphoid, a vicious callus of the radius, or an avascular necrosis of one of the carpal bones.
* In case of failure of medical treatment for at least one year: analgesics of the appropriate level for the pain, NSAIDs, wearing of an analgesic orthosis, rehabilitation by a physiotherapist +/- intra-articular injections of corticoids or hyaluronic acid.
* Informed consent form signed by the patient
* Women of childbearing age must have a negative pregnancy test (serum or urine) (detection threshold (sensitivity): 25 mIU hCG/ml). Patients of both sexes must use reliable contraception.
* Beneficiaries or members of a social security system

Exclusion Criteria:

* Use of antiplatelet drugs, aspirin, anti vitamin K drugs less than 15 days prior to inclusion that may interfere with the quality or therapeutic effect of the investigational drug
* Chronic treatment with oral corticosteroids or less than 2 weeks old
* Intra-articular corticoid injection less than 2 months old
* Intra-articular injection of hyaluronic acid less than 2 months old
* NSAIDs taken less than 15 days ago
* Recent fever or infection (bacterial or viral) less than one month old
* Current or chronic infectious diseases (viral or bacterial) as evidenced by clinical and/or biological elements (inflammatory work-up: VS, CRP, Fibrinogen)
* Autoimmune diseases attested to by questioning, or clinical and/or biological elements (inflammatory workup: VS, CRP, fibrinogen) and which may interfere with the quality or therapeutic effect of the investigational drug
* Inflammatory arthritis
* Microcrystalline arthritis
* History of surgery for the treatment of osteoarthritis of the tested wrist: total denervation of the wrist, resection of the first row of the carpus, arthrodesis, arthroplasty
* Congenital or acquired immune deficiency
* Malignant tumors under treatment or history of malignant tumors less than 5 years old
* Contraindications to MRI: metallic foreign bodies (ferromagnetic material) and metallic implants (pacemakers, heart valves, vascular clips, surgical clips or staples, cochlear implants, any implanted electronic medical material or device (e.g. insulin pump), orthopedic medical prostheses.
* Contraindications to local anesthetics.
* Contraindications to local anesthesia or surgery
* Positive markers for the following active infectious diseases: HIV 1 and HIV 2 human immunodeficiency virus infection; HTLV I infection; Hepatitis B virus infection; Hepatitis C virus infection; Syphilis causative agent infection. (Order of November 4, 2014 on the screening of infectious diseases during autologous therapeutic samples provided for in Article R. 1211-22-1 of the Public Health Code and amending the order of May 14, 2010 setting the content of information allowing the use of human body elements and products for therapeutic purposes)
* Body mass index (BMI) less than 18kg/m2 not allowing to obtain a sufficient quantity of adipose tissue for the manufacturing of the experimental MTI-PP and exposing the patient to a significant discomfort during the liposuction procedure
* Coagulation disorders that may interfere with the quality or therapeutic effect of the investigational drug:
* Thrombocytopenia < 150 G/L
* Thrombocytosis > 450 G/L
* Known thrombopathy
* TP < 70% o Patient/hematopoietic ratio
* Patient to Witness APTT ratio > 1.20
* Anemia < 10g/dl contraindicating peripheral venous blood sampling
* Pregnant or breastfeeding women
* Persons of legal age (under guardianship or trusteeship)
* Persons participating simultaneously in another research project involving the human person or in a period of exclusion from a previous research project
* Persons staying in a health or social institution
* Persons in an emergency situation
* Persons deprived of liberty
* Persons who are not beneficiaries of a social security system
* Absence or refusal to give informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-02-17 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Pain intensity measured on the visual analog scale (EVA) | 6 Months
  The patient will indicate his or her pain using a cross on a 10 cm scale called the VAS score. The VAS is rated from 0 to 100 by the evaluator. The higher the patient's score, the greater the pain.

SECONDARY OUTCOMES:
Pain intensity measured on the visual analog scale (EVA) | Day 7, 3 Months and 1 Year
  The patient will indicate his or her pain using a cross on a 10 cm scale called the VAS score. The VAS is rated from 0 to 100 by the evaluator. The higher the patient's score, the greater the pain.
Combined assessment of function and pain by the PRWE score | 3 Months, 6 Months and 1 Year
  The PRWE (Patient-Rated Wrist Evaluation) is a specific wrist function and pain assessment score. The questionnaire consists of 15 items, 5 of which focus on pain (50 points) and 10 on wrist function (100 points). We will use the combined score in which the total points for wrist function are divided by 2 and added to the pain score to obtain a total score out of 100 points.
Assessment of upper limb function by the DASH score | 3 Months, 6 Months and 1 Year
  The DASH (Disabilities of the Arm, Shoulder and Hand) is a subjective self-assessment questionnaire of the overall functional capacity of both upper limbs. The questionnaire consists of 30 questions covering difficulty with specific activities of daily living, social relationships, and specific symptoms: pain, strength, mobility and sleep. The overall score is presented as a score out of 100 by the following calculation method: [(sum of n responses)-1] x 25n. The score is only valid if 90% of the questions have been filled in by the patient (i.e. 3 missing values at most).
Assessment of wrist strength by dynamometry | 3 Months, 6 Months and 1 Year
  Wrist grip strength will be assessed by the average score of 3 consecutive measurements on the Jamar hydraulic hand dynamometer.
Measurement of wrist joint amplitudes | 3 Months, 6 Months and 1 Year
  The joint amplitudes of the wrist will be measured with a goniometer :
  * in radial tilt
  * in ulnar tilt
  * in flexion
  * in extension These measurements are noted for the wrist with osteoarthritis and the contralateral wrist.
Overall change perceived by the patient | 3 Months, 6 Months and 1 Year
  The patient's overall perceived change will be assessed using the 7-level Likert scale (Check the box that best describes the current condition of your wrist, compared to before the procedure." Much better, Better, Slightly better, No change, Slightly worse, Worse, Much worse).
Patient satisfaction | Day 7, 3 Months
  The patient will answer using the 3-level Likert scale if he/she is satisfied with the therapeutic procedure (Denervation or intra-articular injection of the product under study) ("Check the box that best describes your level of satisfaction with the intervention." (satisfied vs. neither satisfied-nor dissatisfied or dissatisfied; improved vs. no change or worse)The patient will also be asked if he/she would recommend this procedure to a loved one.
MRI evaluation of cartilage lesions in the "study treatment" group | 6 Months
  Pre- and post-operative MRI analysis in the "study treatment" group will allow quantitative assessment of the variation in cartilage relaxation time on gradient echo and 3D high-resolution 3T MRI sequences.

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — Assistance Publique Hôpitaux Marseille; Alice MAYOLY, Principal Investigator — Assistance Publique Hôpitaux Marseille
Locations (1):
- Assistance Publique Hôpitaux Marseille, Marseille, Bouches-du-Rhône, France